CLINICAL TRIAL: NCT03081143
Title: Ramucirumab Plus Irinotecan / Leucovorin / 5-FU Versus Ramucirumab Plus Paclitaxel in Patients with Advanced or Metastatic Adenocarcinoma of the Stomach or Gastroesophageal Junction, Who Failed One Prior Line of Palliative Chemotherapy - the Phase II/III RAMIRIS Study
Brief Title: Ramucirumab Plus FOLFIRI Versus Ramucirumab Plus Paclitaxel in Patients with Advanced or Metastatic Gastric Cancer, Who Failed One Prior Line of Palliative Chemotherapy
Acronym: RAMIRIS
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAMIRIS; AIO-STO-0415 (Other: AIO)
Record Dates: First submitted 2017-03-06; First posted 2017-03-16 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Advanced Gastric or EGJ Cancer
MeSH Terms: interventions — IFL protocol; Ramucirumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FOLFIRI plus Ramucirumab (Experimental): Ramucirumab 8 mg/kg i.v. infusion on day 1 and 15 of a 28-day cycle plus FOLFIRI (Irinotecan 180 mg/m2; i.v. bolus of 5-FU 400 mg/m2, i.v. infusion of leucovorin 400 mg/m2 , followed by a 46-hour continuous administration of 5-FU 2400 mg/m2 on day 1 and 15 of a 28-day cycle)
  Interventions: Drug: FOLFIRI; Drug: Ramucirumab
- Paclitaxel plus Ramucirumab (Active Comparator): Ramucirumab 8 mg/kg i.v. infusion on day 1 and 15 of a 28-day cycle plus Paclitaxel 80 mg/m2 on day 1, 8, 15
  Interventions: Drug: Ramucirumab; Drug: Paclitaxel

INTERVENTIONS:
Drug: FOLFIRI — Irinotecan 180 mg/m2; i.v. bolus of 5-FU 400 mg/m2, i.v. infusion of leucovorin* 400 mg/m2 , followed by a 46-hour continuous administration of 5-FU 2400 mg/m2 on day 1 and 15 of a 28-day cycle
  Arms: FOLFIRI plus Ramucirumab
Drug: Ramucirumab — 8 mg/kg i.v. infusion on day 1 and 15 of a 28-day cycle
Drug: Paclitaxel — 80 mg/m2 on day 1, 8, 15
  Arms: Paclitaxel plus Ramucirumab

SUMMARY:
This clinical trial will evaluate whether it is beneficial in terms of prolongation of survival to combine FOLFIRI (standard treatment) with ramucirumab compared to the standard treatment of ramucirumab plus paclitaxel in patients with advanced gastric cancer after failure of one prior line of palliative chemotherapy. This trial aims to investigate the efficacy and safety of ramucirumab plus FOLFIRI (investigational arm A) compared to paclitaxel plus ramucirumab (control arm B).

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Male or female* ≥ 18 years of age; Patients in reproductive age must be willing to use adequate contraception (that results in a failure rate of <1% per year) during the study and for 3 months after the end of ramucirumab treatment (appropriate contraception is defined as surgical sterilization (e.g. bilateral tubal ligation, vasectomy), hormonal contraception (including oral contraceptive pills (combination of estrogen and progesterone), vaginal ring, injectables, implants, intrauterine devices (IUDs) and intrauterine hormone-releasing system (IUS)), nonhormonal IUDs and complete abstinence). Female patients with childbearing potential need to have a negative pregnancy test within 7 days before study start.
3. Histologically proven gastric adenocarcinoma including adenocarcinoma of the esophagogastric junction
4. Metastatic or locally advanced disease, not amenable to potentially curative resection
5. Phase II only: Documented objective radiological or clinical disease progression during or within 6 months of the last dose of first-line platinum and fluoropyrimidine doublet with or without anthracycline or docetaxel. Neoadjuvant/adjuvant treatment is not counted unless progression occurs <6 months after completion of the treatment. In these cases neoadjuvant/adjuvant treatment is counted as one line.

   OR Phase III only: Radiological or clinical disease progression during or after the last dose of a first-line platinum, fluoropyrimidine-containing therapy. Patients must also have received a taxane with the first-line or during their adjuvant or neoadjuvant therapy or both. Neoadjuvant/adjuvant platinum containing therapy is permitted and is counted as first-line therapy if progression occurs <12 months after completion of the treatment. If progression occurred ≥ 12 months after completion of neoadjuvant/adjuvant therapy, the therapy is not counted as a treatment line. At decision of the investigator, different regimens can be considered as one line of prior treatment, in case these were administrated as a sequential or alternating therapy.
6. Measurable or non-measurable but evaluable disease
7. ECOG performance status 0-1
8. Life expectancy > 12 weeks
9. Adequate hematological, hepatic and renal functions:

   * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
   * Platelets ≥ 100 x 10^9/L
   * Hemoglobin ≥9 g/dL (5.58 mmol/L)
   * Total bilirubin ≤ 1.5 times the upper normal limit (UNL)
   * AST (SGOT) and ALT (SGPT) ≤ 2.5 x UNL in absence of liver metastases, or ≤ 5 x UNL in presence of liver metastases; AP ≤ 5 x UNL
   * Serum creatinine ≤ 1.5 x upper limit of normal, or creatinine clearance (measured via 24-hour urine collection) ≥40 mL/minute (that is, if serum creatinine is >1.5 times the ULN, a 24-hour urine collection to calculate creatinine clearance must be performed)
   * Urinary protein ≤1+ on dipstick or routine urinalysis (UA; if urine dipstick or routine analysis is ≥2+, a 24-hour urine collection for protein must demonstrate <1000 mg of protein in 24 hours to allow participation in this protocol)
   * Adequate coagulation function as defined by International Normalized Ratio (INR) ≤ 1.5, and a partial thromboplastin time (PTT) ≤ 5 seconds above the ULN (unless receiving anticoagulation therapy). Patients receiving warfarin/ phenprocoumon must be switched to low molecular weight heparin and have achieved stable coagulation profile prior to first dose of protocol therapy.
10. Ability to comply with scheduled assessments and with management of toxicities

Exclusion Criteria:

1. Other tumor type than adenocarcinoma (e.g. leiomyosarcoma, lymphoma) or a second cancer except in patients with squamous or basal cell carcinoma of the skin or carcinoma in situ of the cervix that has been effectively treated. Patients curatively treated and disease-free for at least 5 years will be discussed with the sponsor before inclusion
2. Squamous gastric cancer
3. Concurrent chronic systemic immune therapy, chemotherapy, or hormone therapy not indicated in the study protocol
4. Phase II only: Previous therapy with paclitaxel or FOLFIRI Phase III only: Previous therapy with FOLFIRI
5. Current treatment with any anti-cancer therapy ≤ 2 weeks prior to study treatment start unless rapidly progressing disease is measured
6. Concurrent treatment with any other anti-cancer therapy
7. Previous exposure to a VEGF or VEGFR inhibitor or any antiangiogenic agent, or prior enrolment in this study
8. Patient has undergone major surgery within 28 days prior to first dose of protocol therapy, or minor surgery/subcutaneous venous access device placement within 7 days prior to first dose of protocol therapy. The patient has elective or planned major surgery to be performed during the course of the clinical trial
9. Grade 3-4 GI bleeding within 3 months prior to enrollment
10. History of deep vein thrombosis (DVT), pulmonary embolism (PE), or any other significant thromboembolism (venous port or catheter thrombosis or superficial venous thrombosis are not considered "significant") during the 3 months prior to first dose of protocol therapy
11. Cirrhosis at a level of Child-Pugh B (or worse) or cirrhosis (any degree) and a history of hepatic encephalopathy or clinically meaningful ascites resulting from cirrhosis. Clinically meaningful ascites is defined as ascites from cirrhosis requiring diuretics or paracentesis.
12. The patient has uncontrolled known brain or leptomeningeal metastases
13. Known allergic/ hypersensitivity reaction to any of the components of the treatment
14. Contraindications to the use of atropine
15. Other serious illness or medical conditions within the last 12 months prior to study drug administration
16. Any arterial thromboembolic events, including but not limited to myocardial infarction, transient ischemic attack, cerebrovascular accident, or unstable angina, within 6 months prior to first dose of protocol
17. The patient has uncontrolled or poorly-controlled hypertension (>160 mmHg systolic or > 100 mmHg diastolic for >4 weeks) despite standard medical management
18. Active uncontrolled infection
19. Current history of chronic diarrhea
20. Active disseminated intravascular coagulation
21. Any other serious concomitant disease or medical condition that in the judgment of the investigator renders the subject at high risk of treatment complication or reduced the probability of assessing clinical effect
22. Known Dihydropyrimidine dehydrogenase (DPD) deficiency
23. Prior history of GI perforation/fistula (within 6 months of first dose of protocol therapy) or risk factors for perforation.
24. Serious or nonhealing wound, ulcer, or bone fracture within 28 days prior to first dose of protocol therapy
25. The patient is receiving chronic antiplatelet therapy, including aspirin, nonsteroidal anti-inflammatory drugs (NSAIDs, including ibuprofen, naproxen, and others), dipyridamole or clopidogrel, or similar agents. Once-daily aspirin use (maximum dose 325 mg/day) is permitted
26. Concurrent treatment with other experimental drugs or participation in another clinical trial with any investigational drug within 30 days prior to treatment start or at the same time as this study
27. Lack of resolution of all toxic effects (excluding alopecia) of prior chemotherapy, prior radiotherapy or surgical procedure to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) grade < 1. Note: Neuropathy due to prior chemotherapy is allowed if not > NCI Grade II according to CTCAE version 4.03
28. Subject pregnant or breast feeding, or planning to become pregnant within 3 months after the end of treatment
29. Subject (male or female) is not willing to use highly effective methods of contraception (per institutional standardCTFG-Guideline) during treatment and for 3 months (male or female) after the end of treatment
30. Patients known to have a HER 2 positive Cancer who have not been treated already with a HER 2 targeting agent.
31. Patients with a psychiatric illness or patients imprisoned or working in the institution of the treating physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 429 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
OS Rate at 6 months primary endpoint for phase II | 6 months after randomization
  OS Rate at 6 months is defined at the proportion of patients being known to be alive at 6 months after randomisation
overall survival (OS) co-primary endpoint for phase III | from date of randomization to 1 year after end of treatment
  duration from date of randomization to death
Objective Overall Response Rate (ORR) co-primary endpoint for phase III | from randomization for the time of treatment with a maximum of 1 year
  proportion of patients with complete or partial response (CR + PR) according to RECIST 1.1

SECONDARY OUTCOMES:
Progression-free survival | from date of first study drug administration to up to 1 year after study completion
  duration from the first study drug administration to the first documented evidence of disease progression or death
Overall response rate (CR + PR) - endpoint for phase II | from randomization for the time of treatment with a maximum of 1 year
  proportion of patients with complete or partial response (CR + PR) according to RECIST 1.1
Disease control rate (CR + PR + SD) | from randomization for the time of treatment with a maximum of 1 year
  proportion of patients with complete or partial response or stable disease (CR + PR + SD) according to RECIST 1.1
incidence and severity of adverse events according to CTC criteria | from randomization until 30 days after the last dose of study drug
  incidence and severity of adverse events according to CTC criteria
Patient reported outcomes: quality of life according to questionnaire EORTC-QLQ-C30 | from randomization until 30 days after the last dose of study drug
  quality of life scores according to validated questionnaire EORTC-QLQ-C30

CONTACTS AND LOCATIONS:
Overall Officials: Salah-Eddin Al-Batran, Prof, Study Chair — Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest
Locations (16):
- Austria (3):
  - Ordensklinikum Linz GmbH, Barmherzige Schwestern, Linz, Upper Austria
  - Landeskrankenhaus Feldkirch - Rankweil, Rankweil, Vorarlberg
  - Wiener Neustadt, Landesklinikum, Wiener Neustadt
- Germany (12):
  - HELIOS Klinikum Bad Saarow, Bad Saarow
  - Charité - Universitätsmedizin Berlin, Berlin
  - HELIOS Klinikum Berlin Buch, Berlin
  - Klinikum Bielefeld Mitte, Bielefeld
  - Kliniken Essen Mitte, Essen
  - Krankenhaus Nordwest, Frankfurt
  - Hämatologisch-Onkologische Praxis Eppendorf (HOPE), Hamburg
  - Ortenau Klinikum, Lahr
  - Universitäres Krebszentrum Leipzig, Leipzig
  - Technische Universität München, München
  - Universitätsklinikum Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm
- U.O. Oncologia Medica, Università Cattolica Sacro Cuore, Rome, Italy

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared.

REFERENCES:
- [Background] Lorenzen S, Thuss-Patience P, Pauligk C, Gokkurt E, Ettrich T, Lordick F, Stahl M, Reichardt P, Sokler M, Pink D, Probst S, Hinke A, Goetze TO, Al-Batran SE. FOLFIRI plus ramucirumab versus paclitaxel plus ramucirumab as second-line therapy for patients with advanced or metastatic gastroesophageal adenocarcinoma with or without prior docetaxel - results from the phase II RAMIRIS Study of the German Gastric Cancer Study Group at AIO. Eur J Cancer. 2022 Apr;165:48-57. doi: 10.1016/j.ejca.2022.01.015. Epub 2022 Feb 21. PMID 35202974
- [Derived] Lorenzen S, Schwarz A, Pauligk C, Goekkurt E, Stocker G, Knorrenschild JR, Illerhaus G, Dechow T, Moehler M, Moulin JC, Pink D, Stahl M, Schaaf M, Goetze TO, Al-Batran SE. Ramucirumab plus irinotecan / leucovorin / 5-FU versus ramucirumab plus paclitaxel in patients with advanced or metastatic adenocarcinoma of the stomach or gastroesophageal junction, who failed one prior line of palliative chemotherapy: the phase II/III RAMIRIS study (AIO-STO-0415). BMC Cancer. 2023 Jun 19;23(1):561. doi: 10.1186/s12885-023-11004-z. PMID 37337155